CLINICAL TRIAL: NCT04591080
Title: A Comparison Between TiNbTaZr (GUMMETAL) and Stainless-steel Alloy for Space Closure With Sliding Mechanics A Pilot Randomized Clinical Trial
Brief Title: A Comparison Between GUMMETAL and SS Orthodontic Wires in Space Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Lubomyr Ravlyk, Orthodontic Resident, State University of New York at Buffalo
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: GMTSS
Record Dates: First submitted 2020-10-11; First posted 2020-10-19 (Actual); Results first posted 2024-04-19 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Malocclusion, Angle Class I
MeSH Terms: conditions — Malocclusion, Angle Class I

STUDY DESIGN:
Intervention Model Description: Split mouth design where one side of the mouth will be receiving the intervention and the other side of the mouth the control treatment.
Who Masked: Participant
Masking Description: The participants will not know which intervention is on which side of their mouth, but will know that they are getting both types of interventions simultaneously, given the split-mouth design of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- GUMMETAL TiNbTaZr (Experimental): TiNbTaZr (Beta-Titanium) Alloy used to manufacture orthodontic archwires. We will be using an archwire with the size of 0.016 x 0.022"
  Interventions: Device: GUMMETAL Orthodontic Wire
- Stainless Steel (CrNi) (Active Comparator): Stainless steel (18% Chromium and 8% Nickel) used as the control, and linked anteriorly to the GUMMETAL counterpart. Size of archwire is 0.016 x 0.022"
  Interventions: Device: Stainless Steel (CrNi)

INTERVENTIONS:
Device: GUMMETAL Orthodontic Wire — Orthodontic archwire made of TiNbTaZr alloy.
  Other Names: TiNbTaZr, Titanium-niobium, Beta-titanium,
  Arms: GUMMETAL TiNbTaZr
Device: Stainless Steel (CrNi) — Stainless steel (18% Chromium and 8% Nickel) used as the control, and linked anteriorly to the GUMMETAL counterpart. Size of archwire is 0.016 x 0.022"
  Arms: Stainless Steel (CrNi)

SUMMARY:
When there is space present between our teeth orthodontically we have the ability to close them through many methods. Using braces as our treatment modality this study will be investigating how efficient a new orthodontic wire is in closing tooth space. This new material is trade-named GUMMETAL and claims to have many benefits to treating patients orthodontically. We will be exploring its efficiency in space closure compared to an industry standard (stainless steel). We predict that the stainless-steel orthodontic wire will be more efficient at space closure than the new GUMMETAL wires.

DETAILED DESCRIPTION:
This will be a randomized pilot split-mouth clinical trial of patients with spaces ≥ 3mm distal to the maxillary canines in need of closure through sliding mechanics. The sample consists of adolescent patients regardless of Angle's molar malocclusion who are receiving comprehensive full fixed appliance orthodontic treatment. Preformed conjoint archwires half being GUMMETAL and the other half SS, will be utilized. Each patient will have one side of the maxilla randomly allocated into the SS or GUMMETAL treatment group. The study will follow a split-mouth design to reduce the confounding variables from patient to patient on space closure mechanics. The maxillary arch in each subject will be randomized into a SS side or GM side using a random number generator. Spaces will be measured at; T0 is initial records, T1 is initiation of space closure, T2 will be 4 weeks after the initiation of space closure, T3 is another 4 weeks of space closure evaluation and T4 will be the final evaluation of space closure after 4 weeks from T3, via 3D intraoral scans of maxillary arches. Space measurement and calculations will utilize 3Shape software to measure the distance of canine movement based off the distal surface. Sliding mechanics will be activated through NiTi coil springs from the maxillary canines to the maxillary molars. The force will be standardized to 150 gms and will be measured each visit. The same provider will activate the NiTi coil spring for retraction, along with data collection. Superimposition of scans will be utilized to assess outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Full permanent dentition (except third molars)
* Good general and oral health
* Bilateral spaces 3 >/= mm distal to the maxillary canines
* Normal and hypodivergent growth pattern
* Any dental malocclusion
* Good Oral Hygiene

Exclusion Criteria:

* Systemic diseases or syndrome
* Abnormalities in teeth size and/or shape
* Previous orthodontic treatment
* Anti-inflammatory medication
* Craniofacial anomalies
* Hyperdivergent growth pattern
* Periodontal disease / attachment loss exceeding 25% of root length
* Significant pre or in-treatment root resorption

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thikriat Al-Jewair, Study Chair — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
We will not be sharing any IPD information with any other researchers.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a split-mouth pilot study.
  A total of 12 participants were enrolled. 24 adult canine teeth were randomized 1:1 to the control and intervention conditions (sides Rt vs Lt) resulting in 12 canines receiving the control treatment and 12 canines receiving the intervention.
  A total of 6 participants completed the study.6 canines receiving the control treatment and 6 canines receiving the intervention.
Units Other Than Participants: Right vs left canine
Groups:
- Control: Control: Stainless steel (18% Chromium and 8% Nickel) used as the control, and linked anteriorly to the GUMMETAL counterpart. Size of archwire is 0.016 x 0.022". Stainless Steel (CrNi): Stainless steel (18% Chromium and 8% Nickel) used as the control, and linked anteriorly to the GUMMETAL counterpart. Size of archwire is 0.016 x 0.022"
- Intervention: This is a split-mouth study. Each subject was allocated to both the control and intervention groups. The unit of assessment is the right and left maxillary canine teeth.
  Intervention: TiNbTaZr (Beta-Titanium) Alloy used to manufacture orthodontic archwires. We will be using an archwire with the size of 0.016 x 0.022". GUMMETAL Orthodontic Wire: Orthodontic archwire made of TiNbTaZr alloy.
Period: Overall Study
Arm/Group | Control | Intervention
Started | 12; 12 Right vs left canine | 12; 12 Right vs left canine
Completed | 6; 6 Right vs left canine | 6; 6 Right vs left canine
Not Completed | 6; 6 Right vs left canine | 6; 6 Right vs left canine

BASELINE CHARACTERISTICS:
Groups:
- All Participants: This is a split-mouth study. Each subject was allocated to both the control and intervention groups. The unit of assessment is the right and left maxillary canine teeth.
  Intervention: TiNbTaZr (Beta-Titanium) Alloy used to manufacture orthodontic archwires. We will be using an archwire with the size of 0.016 x 0.022". GUMMETAL Orthodontic Wire: Orthodontic archwire made of TiNbTaZr alloy.
  Control: Stainless steel (18% Chromium and 8% Nickel) used as the control, and linked anteriorly to the GUMMETAL counterpart. Size of archwire is 0.016 x 0.022". Stainless Steel (CrNi): Stainless steel (18% Chromium and 8% Nickel) used as the control, and linked anteriorly to the GUMMETAL counterpart. Size of archwire is 0.016 x 0.022"
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Total Amount of Canine Retraction
Description: Canine movement measured at distal marginal ridge
Time Frame: 12 weeks
Population: 2 canine teeth were assessed per subject (total of 6 subjects completed the study)
Measure: Median (Inter-Quartile Range); unit: mm
Units Other Than Participants: Canine teeth
Arm/Group | GUMMETAL TiNbTaZr | Stainless Steel (CrNi)
Number analyzed (Participants) | 6 | 6
Number analyzed (Canine teeth) | 12 | 12
mm | 3.41 [2.10 to 4.76] | 3.71 [1.62 to 6.45]

2. Secondary Outcome: 3-Dimensional Control of Canine Movement Assessment
Description: Canine position (tip, rotation, angulation) will be assessed from initial to final position
Time Frame: 12 weeks
Population: 2 canine teeth per subject
Measure: Median (Inter-Quartile Range); unit: degrees
Units Other Than Participants: Canine teeth
Arm/Group | GUMMETAL TiNbTaZr | Stainless Steel (CrNi)
Number analyzed (Participants) | 6 | 6
Number analyzed (Canine teeth) | 12 | 12
degrees | 7.90 [6.74 to 8.99] | 7.25 [6.71 to 8.16]

3. Secondary Outcome: Rate of Canine Retraction Per Month
Description: Rate of canine retraction in mm per month
Time Frame: 12 weeks
Population: 2 canine teeth per subject
Measure: Median (Inter-Quartile Range); unit: mm/month
Units Other Than Participants: Canine teeth
Arm/Group | GUMMETAL TiNbTaZr | Stainless Steel (CrNi)
Number analyzed (Participants) | 6 | 6
Number analyzed (Canine teeth) | 12 | 12
mm/month | 1.14 [0.69 to 1.59] | 1.42 [0.54 to 2.15]

ADVERSE EVENTS:
Time Frame: Throughout study completion: An average of 6 months
Description: No risks anticipated
Groups:
- All Participants: This is a split-mouth study: Each person was allocated a control and intervention sides (Right vs left maxillary canines).
  Stainless steel (18% Chromium and 8% Nickel) used as the control, and linked anteriorly to the GUMMETAL counterpart. Size of archwire is 0.016 x 0.022"
  TiNbTaZr (Beta-Titanium) Alloy size of 0.016 x 0.022" was used as the intervention.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT04591080/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-12): https://cdn.clinicaltrials.gov/large-docs/80/NCT04591080/ICF_001.pdf